CLINICAL TRIAL: NCT00535782
Title: A Mechanism of Action Study to Evaluate the Effects of IL-6 Receptor Blockade With Tocilizumab (TCZ) on Lipids, Arterial Stiffness, and Markers of Atherogenic Risk in Patients With Moderate to Severe Active Rheumatoid Arthritis (RA).
Brief Title: A Study of the Effect of Tocilizumab on Markers of Atherogenic Risk in Patients With Moderate to Severe Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WA19923; 2007-001114-17
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Results first posted 2012-11-14 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- TCZ + MTX (Experimental): Participants received 8 mg/kg tocilizumab (TCZ) by intravenous infusion (IV) every 4 weeks plus methotrexate (MTX) 7.5-25 mg (oral or parenteral) weekly for the first 24 weeks. From Week 24 to Week 104, participants received open-label TCZ 8 mg/kg every 4 weeks plus 7.5-25 mg MTX weekly.
  Interventions: Drug: Tocilizumab; Drug: Methotrexate
- Placebo + MTX (Placebo Comparator): Participants received placebo intravenous infusion (IV) every 4 weeks plus methotrexate (MTX) 7.5-25 mg (oral or parenteral) weekly for the first 24 weeks. From Week 24 to 104, participants received open-label tocilizumab (TCZ) 8 mg/kg every 4 weeks plus 7.5-25 mg MTX.
  Interventions: Drug: Tocilizumab; Drug: Placebo; Drug: Methotrexate

INTERVENTIONS:
Drug: Tocilizumab — Administered by intravenous infusion, 8 mg/kg every 4 weeks.
  Other Names: RoActemra; Actemra
Drug: Placebo — Placebo to tocilizumab administered by intravenous infusion every 4 weeks.
  Arms: Placebo + MTX
Drug: Methotrexate — Administered orally or parenterally, 7.5-25 mg weekly.

SUMMARY:
This 2 arm study will investigate the effects of tocilizumab on lipids, arterial stiffness, and markers of atherogenic risk in patients with moderate to severe active rheumatoid arthritis. In Part 1 of the study, patients will be randomized to receive either tocilizumab 8mg/kg intravenously or placebo every 4 weeks, in combination with methotrexate 7.5-25 mg weekly. In Part 2, all patients will receive open-label treatment with tocilizumab plus methotrexate.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-75 years of age
* rheumatoid arthritis (RA) of >6 months duration
* able to receive outpatient treatment
* on methotrexate for at least 12 weeks before entering study, at a stable dose of 7.5-25 mg/week for the last 8 weeks
* oral corticosteroids and non-steroidal anti-inflammatory drugs (NSAIDS) permitted, if at a stable dose for 4 weeks before study start

Exclusion Criteria

* major surgery (including joint surgery) within 8 weeks prior to screening, or planned surgery within 6 months after entering study
* history of, or current inflammatory joint disease or rheumatic autoimmune disease other than RA
* inadequate response to anti-tumor necrosis factor (TNF) agent during the 6 months prior to baseline, or inadequate response to >2 anti-TNF agents
* initiation of treatment with lipid lowering agents within 12 weeks prior to baseline

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2007-10-31 (Actual); Primary Completion 2008-09-30 (Actual); Study Completion 2011-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (40):
- United States (26):
  - Pinnacle Research Group; Llc, Central, Anniston, Alabama
  - Rheumatology Associates of North Alabama, Huntsville, Alabama
  - Advanced Arthritis Care & Research, Scottsdale, Arizona
  - Catalina Pointe Clinical Research, Inc., Tucson, Arizona
  - Pacific Arthritis Care Center, Los Angeles, California
  - Arthritis & Rheumatism; Disease Specialities, Aventura, Florida
  - Science and Research Institute, Inc., Jupiter, Florida
  - Arthritis Center Palm Harbor, Palm Harbor, Florida
  - Arthritis Rsrch of Florida, Inc., Palm Harbor, Florida
  - Sarasota Arthritis Center; Research Dept, Sarasota, Florida
  - Burnette & Silverfield, MDS, Tampa, Florida
  - Arthritis & Rheumatology of Georgia, Atlanta, Georgia
  - Deerbrook Medical Associates, Vernon Hills, Illinois
  - Johns Hopkins Uni, Baltimore, Maryland
  - Borgess Research Institute, Kalamazoo, Michigan
  - Jackson Arthritis Clinic, Flowood, Mississippi
  - Physicians Group, LC DBA Rheumatology & Internal Medicine Associates, St Louis, Missouri
  - NJP Clinical Research, Clifton, New Jersey
  - Asheville Arthritis & Osteoporosis Center, PA, Asheville, North Carolina
  - Health Research of Oklahoma, Llc, Oklahoma City, Oklahoma
  - Lehigh Valley Hospital; Dept of Medicine, Allentown, Pennsylvania
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - Clinical Research Center of Reading, Wyomissing, Pennsylvania
  - Houston Inst. For Clinical Research, Houston, Texas
  - Texas Research Center, Sugar Land, Texas
  - South Puget Sound Clinical Research, Olympia, Washington
- Canada (10):
  - The Governors of the Uni of Alberta; Heritage Medical Research Centre, Edmonton, Alberta
  - Laurel Medical Clinic, Vancouver, British Columbia
  - Manitoba Clinic, Winnipeg, Manitoba
  - Nexus Clinical Research Centre, St. John's, Newfoundland and Labrador
  - Dr. William G. Bensen Medicine Professional Corporation, Hamilton, Ontario
  - Credit Valley, Rheumatology, Mississauga, Ontario
  - Rheumatology Research Associates, Ottawa, Ontario
  - Private Practice, Toronto, Ontario
  - Chus Hopital Fleurimont, Sherbrooke, Quebec
  - Centre Re Recherche Saint-Louis, Québec
- Ponce School of Medicine; Caimed Center, Ponce, Puerto Rico
- United Kingdom (3):
  - Glasgow Royal Infirmary; Centre For Rheumatic Diseases, Glasgow
  - Trafford General Hospital; Rheumatology, Manchester
  - Royal Victoria Infirmary; Clinical Research Facility, Newcastle upon Tyne

REFERENCES:
- [Derived] Wang J, Bansal AT, Martin M, Germer S, Benayed R, Essioux L, Lee JS, Begovich A, Hemmings A, Kenwright A, Taylor KE, Upmanyu R, Cutler P, Harari O, Marchini J, Criswell LA, Platt A. Genome-wide association analysis implicates the involvement of eight loci with response to tocilizumab for the treatment of rheumatoid arthritis. Pharmacogenomics J. 2013 Jun;13(3):235-41. doi: 10.1038/tpj.2012.8. Epub 2012 Apr 10. PMID 22491018

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1: TCZ + MTX: During Part 1 of the study participants in this group received 8 mg/kg tocilizumab (TCZ) by intravenous infusion (IV) every 4 weeks plus methotrexate (MTX) 7.5-25 mg (oral or parenteral) weekly for 24 weeks.
- Part 1: Placebo + MTX: During Part 1 of the study participants in this group received placebo intravenous infusion (IV) every 4 weeks plus methotrexate (MTX) 7.5-25 mg (oral or parenteral) weekly for 24 weeks.
- Part 2: TCZ + MTX: During Part 2 of the study, from Week 24 to Week 104, all participants received 8 mg/kg tocilizumab (TCZ) by intravenous infusion (IV) every 4 weeks plus methotrexate (MTX) 7.5-25 mg (oral or parenteral) weekly.
Period: Part 1: 24-Week Double-blind Period
Arm/Group | Part 1: TCZ + MTX | Part 1: Placebo + MTX | Part 2: TCZ + MTX
Started | 69 | 63 | 0
Treated With TCZ + MTX | 69 | 2 (1 misrandomized patient received the TCZ in error, and 1 patient received TCZ as rescue therapy.) | 0
Treated With Placebo + MTX | 0 | 62 | 0
Completed | 65 | 59 | 0
Not Completed | 4 | 4 | 0
Period: Part 2: 80-Week Open-label Period
Arm/Group | Part 1: TCZ + MTX | Part 1: Placebo + MTX | Part 2: TCZ + MTX
Started | 0 | 0 | 124
Completed | 0 | 0 | 98
Not Completed | 0 | 0 | 26

BASELINE CHARACTERISTICS:
Groups:
- TCZ + MTX: During Part 1 of the study participants received 8 mg/kg tocilizumab (TCZ) by intravenous (IV) infusion every 4 weeks plus methotrexate (MTX) 7.5-25 mg (oral or parenteral) weekly for 24 weeks. During Part 2, from Week 24 to Week 104, participants received open-label 8 mg/kg TCZ every 4 weeks plus 7.5-25 mg MTX weekly.
- Placebo + MTX: During Part 1 of the study participants received placebo intravenous (IV) infusion every 4 weeks plus methotrexate (MTX) 7.5-25 mg (oral or parenteral) weekly for 24 weeks. During Part 2, from Week 24 to Week 104, participants received 8 mg/kg TCZ IV every 4 weeks plus 7.5-25 mg MTX weekly.
- Total: Total of all reporting groups
Arm/Group | TCZ + MTX | Placebo + MTX | Total
Number analyzed (Participants) | 69 | 63 | 132
Age, Customized [Number; unit: participants]
  <52 years | 23 | 20 | 43
  ≥52 years | 46 | 43 | 89
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 47 | 104
  Male | 12 | 16 | 28
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1 | 3 | 4
  Black | 2 | 4 | 6
  Other | 3 | 1 | 4
  White | 63 | 55 | 118
Region of Enrollment [Number; unit: participants]
  United States | 41 | 46 | 87
  Canada | 23 | 16 | 39
  United Kingdom | 5 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Small Low Density Lipoprotein (sLDL) Particle Numbers
Description: Small LDL particles are associated with an increased risk of cardiovascular disease: more of these small particles lead to a greater risk. The concentration of fasting small LDL particles was determined using the Nuclear Magnetic Resonance (NMR) methodology.
Time Frame: Baseline and Week 12
Population: Intent to treat (ITT) population. All randomized patients who received any part of an infusion of study medication are included. Patients who received an incorrect therapy from that intended are summarized in the group according to the intended randomized treatment group. Last observation carried forward (LOCF) imputation was used.
Measure: Mean (Standard Deviation); unit: nmol/L
Groups:
- TCZ + MTX: Participants received 8 mg/kg tocilizumab (TCZ) by intravenous infusion (IV) every 4 weeks plus 7.5-25 mg of methotrexate (MTX) weekly for the first 24 weeks.
- Placebo + MTX: Participants received placebo intravenous infusion (IV) every 4 weeks plus methotrexate (MTX) 7.5-25 mg (oral or parenteral) weekly for the first 24 weeks.
Arm/Group | TCZ + MTX | Placebo + MTX
Number analyzed (Participants) | 69 | 63
nmol/L
  Baseline (n=63, 59) | 737.79 (467.097) | 792.78 (392.051)
  Week 12 (n=69, 63) | 768.04 (628.281) | 777.71 (394.527)
  Change from Baseline at Week 12 (n=63, 59) | 23.73 (368.273) | 22.41 (237.476)

2. Secondary Outcome: Change From Baseline to Week 24 in Small Low Density Lipoprotein (sLDL) Particle Numbers
Description: as for outcome 1
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | TCZ + MTX | Placebo + MTX
Number analyzed (Participants) | 69 | 63
nmol/L
  Baseline (n=63, 59) | 737.79 (467.097) | 792.78 (392.051)
  Week 24 (n=69, 63) | 792.78 (605.485) | 801.78 (398.910)
  Change from Baseline at Week 24 (n=63, 59) | 39.03 (367.786) | 32.41 (250.576)

3. Secondary Outcome: Change From Baseline to Week 24 in Aortic Pulse Wave Velocity (PWV)
Description: Aortic (central) arterial stiffness was assessed with Pulse Wave Analysis (PWA) of the radial artery and carotid-femoral PWV using applanation tonometry after the patient had rested in a supine position for at least 10 minutes.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | TCZ + MTX | Placebo + MTX
Number analyzed (Participants) | 69 | 63
meters/second
  Baseline (n=69, 59) | 8.97 (1.970) | 9.01 (2.519)
  Week 24 (n=69, 62) | 8.98 (2.337) | 8.85 (2.014)
  Change from Baseline at Week 24 (n=69, 59) | 0.01 (1.946) | -0.20 (1.792)

4. Secondary Outcome: Number of Participants Experiencing Adverse Events (AEs)
Description: A severe AE is an event in which the intensity of the event results in an inability to work or perform normal daily activity.
  A Serious AE is fatal, life-threatening, requires in-patient hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant or requires intervention to prevent one of the above outcomes.
  AEs of special interest include infection, gastrointestinal, infusion reaction (occurring during or within 24 hours of infusion), hepatic disorder, myocardial infarction and stroke.
Time Frame: Up to Week 24
Population: The safety population includes all patients who received any part of an infusion of study drug and who provided at least one assessment of safety. Randomized patients who received the incorrect therapy from that intended are summarized in the group according to the therapy actually received.
Measure: Number; unit: participants
Arm/Group | TCZ + MTX | Placebo + MTX
Number analyzed (Participants) | 70 | 62
participants
  Any AE | 59 | 45
  Severe AE | 7 | 4
  Serious AE | 3 | 2
  Deaths | 0 | 0
  Withdrawals due to AE | 2 | 1
  Pregnancy | 0 | 0
  Infection AEs | 42 | 17
  Gastrointestinal AEs | 22 | 10
  Infusion reaction AEs | 12 | 7
  Hepatic disorder AEs | 0 | 0
  Myocardial infarction | 0 | 0
  Stroke | 0 | 0

5. Primary Outcome: Change From Baseline to Week 12 in Aortic Pulse Wave Velocity (PWV)
Description: as for outcome 3
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | TCZ + MTX | Placebo + MTX
Number analyzed (Participants) | 69 | 63
meters/second
  Baseline (n=69, 59) | 8.97 (1.970) | 9.01 (2.519)
  Week 12 (n=69, 62) | 8.94 (2.510) | 8.39 (1.836)
  Change from Baseline at Week 12 (n=69, 59) | -0.03 (1.970) | -0.68 (1.741)

ADVERSE EVENTS:
Groups:
- All TCZ + MTX: Includes patients who received at least one dose of active tocilizumab (TCZ) regardless of when they received it during the study and whether it was double-blind (Part 1) or open-label (Part 2). Participants received 8 mg/kg TCZ by intravenous infusion (IV) every 4 weeks plus methotrexate (MTX) 7.5-25 mg (oral or parenteral) weekly.
Arm/Group | Part 1: TCZ + MTX | Part 1: Placebo + MTX | All TCZ + MTX
Serious Adverse Events (participants affected / at risk) | 3/70 | 2/62 | 30/130
Other Adverse Events (participants affected / at risk) | 59/70 | 44/62 | 124/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: TCZ + MTX (N=70) | Part 1: Placebo + MTX (N=62) | All TCZ + MTX (N=130)
Arthritis bacterial (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 1
Pneumonia streptococcal (Infections and infestations) | 0 | 0 | 1
Puncture site abscess (Infections and infestations) | 0 | 0 | 1
Staphylococcal abscess (Infections and infestations) | 0 | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 4
Stress cardiomyopathy (Cardiac disorders) | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Multiple drug overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 2
Chest pain (General disorders) | 0 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic artery aneurysm (Hepatobiliary disorders) | 0 | 0 | 1
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1
Sarcoidosis (Immune system disorders) | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Bipolar disorder (Psychiatric disorders) | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1
Aortic stenosis (Vascular disorders) | 0 | 0 | 1
Shock haemorrhagic (Vascular disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Goitre (Endocrine disorders) | 0 | 0 | 1
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: TCZ + MTX (N=70) | Part 1: Placebo + MTX (N=62) | All TCZ + MTX (N=130)
Upper respiratory tract infection (Infections and infestations) | 8 | 6 | 39
Urinary tract infection (Infections and infestations) | 7 | 2 | 25
Bronchitis (Infections and infestations) | 3 | 2 | 23
Sinusitis (Infections and infestations) | 4 | 1 | 19
Nasopharyngitis (Infections and infestations) | 5 | 0 | 16
Gastroenteritis (Infections and infestations) | 1 | 2 | 9
Pneumonia (Infections and infestations) | 0 | 0 | 7
Cellulitis (Infections and infestations) | 1 | 0 | 6
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 6
Lower respiratory tract infection (Infections and infestations) | 2 | 0 | 6
Oral herpes (Infections and infestations) | 1 | 0 | 6
Otitis media (Infections and infestations) | 0 | 0 | 5
Influenza (Infections and infestations) | 1 | 2 | 4
Cystitis (Infections and infestations) | 2 | 0 | 3
Eye infection (Infections and infestations) | 0 | 0 | 3
Laryngitis (Infections and infestations) | 0 | 0 | 3
Localised infection (Infections and infestations) | 1 | 1 | 3
Paronychia (Infections and infestations) | 1 | 0 | 3
Ear infection (Infections and infestations) | 1 | 0 | 2
Folliculitis (Infections and infestations) | 1 | 0 | 2
Furuncle (Infections and infestations) | 1 | 0 | 2
Herpes zoster (Infections and infestations) | 0 | 0 | 2
Infected bites (Infections and infestations) | 1 | 0 | 2
Labyrinthitis (Infections and infestations) | 1 | 0 | 2
Tinea pedis (Infections and infestations) | 0 | 1 | 2
Tooth abscess (Infections and infestations) | 0 | 1 | 2
Viral infection (Infections and infestations) | 0 | 1 | 2
Alveolar osteitis (Infections and infestations) | 0 | 0 | 1
Blister infected (Infections and infestations) | 0 | 0 | 1
Bronchiectasis (Infections and infestations) | 0 | 0 | 1
Burn infection (Infections and infestations) | 0 | 0 | 1
Clostridial infection (Infections and infestations) | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1
Fungal infection (Infections and infestations) | 0 | 1 | 1
Fungal skin infection (Infections and infestations) | 1 | 0 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 1
Gingival infection (Infections and infestations) | 0 | 0 | 1
Helicobacter gastritis (Infections and infestations) | 0 | 0 | 1
Helicobacter infection (Infections and infestations) | 0 | 0 | 1
Hordeolum (Infections and infestations) | 1 | 1 | 1
Impetigo (Infections and infestations) | 0 | 0 | 1
Infected cyst (Infections and infestations) | 0 | 0 | 1
Kidney infection (Infections and infestations) | 0 | 0 | 1
Nail infection (Infections and infestations) | 0 | 0 | 1
Onychomycosis (Infections and infestations) | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 0 | 1
Papilloma viral infection (Infections and infestations) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Rhinitis (Infections and infestations) | 1 | 0 | 1
Sinobronchitis (Infections and infestations) | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 0 | 1
Tinea cruris (Infections and infestations) | 1 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 1
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0 | 1
Wound infection (Infections and infestations) | 0 | 0 | 1
Genital herpes (Infections and infestations) | 1 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 4 | 6 | 16
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 11
Bursitis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 9
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 8
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 6
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 5
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 5
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 4
Rheumatoid nodule (Musculoskeletal and connective tissue disorders) | 2 | 1 | 4
Tendonitis (Musculoskeletal and connective tissue disorders) | 3 | 1 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Bunion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Ligament disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Plantar fascitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 9 | 2 | 22
Nausea (Gastrointestinal disorders) | 1 | 2 | 12
Vomiting (Gastrointestinal disorders) | 4 | 1 | 10
Gastritis (Gastrointestinal disorders) | 5 | 0 | 8
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 7
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 7
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 7
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 6
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 5
Constipation (Gastrointestinal disorders) | 1 | 0 | 5
Mouth ulceration (Gastrointestinal disorders) | 4 | 0 | 5
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 0 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 3
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 3
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 2
Dental caries (Gastrointestinal disorders) | 0 | 0 | 2
Flatulence (Gastrointestinal disorders) | 0 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 1
Barrett's Oesophagus (Gastrointestinal disorders) | 0 | 0 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 1
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Gingivitis (Gastrointestinal disorders) | 1 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 1
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 1
Oesophageal irritation (Gastrointestinal disorders) | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1
Parotid gland enlargement (Gastrointestinal disorders) | 0 | 0 | 1
Peptic ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Periodontitis (Gastrointestinal disorders) | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Stomach discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Oropharnygeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 11
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 4
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 2 | 14
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 1 | 7
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 4
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 1 | 1 | 3
Pruritis (Skin and subcutaneous tissue disorders) | 1 | 1 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Granuloma annulare (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Skin plaque (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 2 | 0 | 8
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 6
Fall (Injury, poisoning and procedural complications) | 1 | 2 | 6
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 4
Joint sprain (Injury, poisoning and procedural complications) | 0 | 1 | 3
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 0 | 3
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 2
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 2
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 2
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 1
Animal scratch (Injury, poisoning and procedural complications) | 0 | 0 | 1
Avulsion fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Incision site haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Muscle injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 2 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural headache (Injury, poisoning and procedural complications) | 1 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fatigue (General disorders) | 2 | 7 | 11
Oedema peripheral (General disorders) | 1 | 0 | 8
Chest pain (General disorders) | 0 | 0 | 4
Pyrexia (General disorders) | 1 | 0 | 4
Influenza like illness (General disorders) | 0 | 1 | 3
Cyst (General disorders) | 1 | 0 | 2
Infusion related reaction (General disorders) | 1 | 0 | 2
Non-cardiac chest pain (General disorders) | 2 | 0 | 2
Chills (General disorders) | 0 | 0 | 1
Feeling hot (General disorders) | 0 | 0 | 1
Impaired healing (General disorders) | 0 | 0 | 1
Infusion site rash (General disorders) | 1 | 0 | 1
Metaplasia (General disorders) | 0 | 0 | 1
Oedema (General disorders) | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 4 | 0 | 15
Dizziness (Nervous system disorders) | 2 | 1 | 9
Amnesia (Nervous system disorders) | 1 | 0 | 2
Migraine (Nervous system disorders) | 1 | 0 | 2
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 2
Aphasia (Nervous system disorders) | 0 | 0 | 1
Carotid artery disease (Nervous system disorders) | 0 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 1
Cauda equina syndrome (Nervous system disorders) | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1
Lethargy (Nervous system disorders) | 1 | 0 | 1
Nerve compression (Nervous system disorders) | 0 | 0 | 1
Tarsal tunnel syndrome (Nervous system disorders) | 0 | 0 | 1
Tremor (Nervous system disorders) | 1 | 0 | 1
Lumbar radiculopathy (Nervous system disorders) | 0 | 1 | 0
Sinus headache (Nervous system disorders) | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 1 | 6
Alanine aminotransferase increased (Investigations) | 0 | 0 | 4
Cardiac murmur (Investigations) | 0 | 0 | 3
Transaminases increased (Investigations) | 1 | 0 | 3
Weight increased (Investigations) | 0 | 0 | 3
Aspartate amniotransferase increased (Investigations) | 0 | 0 | 1
Blood cholesterol increased (Investigations) | 0 | 0 | 1
Blood thyroid stimulating hormone decreased (Investigations) | 0 | 0 | 1
Blood triglycerides increased (Investigations) | 1 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 1
Helicobacter test positive (Investigations) | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 1
Serum ferritin decreased (Investigations) | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 1
Band neutrophil count increased (Investigations) | 0 | 1 | 0
Helicobacter pylori identification test positive (Investigations) | 1 | 0 | 0
Occult blood (Investigations) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 12
Aortic aneurysm (Vascular disorders) | 0 | 0 | 3
Arteriosclerosis (Vascular disorders) | 0 | 1 | 2
Accelerated hypertension (Vascular disorders) | 0 | 0 | 1
Flushing (Vascular disorders) | 1 | 1 | 1
Hot flush (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1
Peripheral artery aneurysm (Vascular disorders) | 0 | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 1
Iliac artery stenosis (Vascular disorders) | 0 | 1 | 0
Phlebitis (Vascular disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 3
Dry eye (Eye disorders) | 1 | 0 | 3
Ocular hyperaemia (Eye disorders) | 0 | 0 | 2
Asthenopia (Eye disorders) | 0 | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 1 | 1 | 1
Conjunctivitis allergic (Eye disorders) | 1 | 0 | 1
Eye irritation (Eye disorders) | 0 | 1 | 1
Eye swelling (Eye disorders) | 0 | 0 | 1
Eyelid cyst (Eye disorders) | 1 | 0 | 1
Glaucoma (Eye disorders) | 1 | 0 | 1
Macular oedema (Eye disorders) | 1 | 0 | 1
Posterior capsule opacification (Eye disorders) | 0 | 0 | 1
Retinal tear (Eye disorders) | 0 | 0 | 1
Ulcerative keratitis (Eye disorders) | 0 | 0 | 1
Visual impairment (Eye disorders) | 0 | 0 | 1
Vitreous floaters (Eye disorders) | 0 | 0 | 1
Myodesopsia (Eye disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 9
Depression (Psychiatric disorders) | 0 | 4 | 5
Anxiety (Psychiatric disorders) | 0 | 1 | 2
Confusional state (Psychiatric disorders) | 1 | 0 | 1
Libido increased (Psychiatric disorders) | 1 | 0 | 1
Restlessness (Psychiatric disorders) | 1 | 0 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 5
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 4
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 1 | 3
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 2
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 6
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 3
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 3
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 2
Lymph node calcification (Blood and lymphatic system disorders) | 0 | 0 | 1
Splenic lesion (Blood and lymphatic system disorders) | 0 | 0 | 1
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 2
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1
Breast calcifications (Reproductive system and breast disorders) | 0 | 0 | 1
Breast cyst (Reproductive system and breast disorders) | 0 | 0 | 1
Breast tenderness (Reproductive system and breast disorders) | 0 | 0 | 1
Genital ulceration (Reproductive system and breast disorders) | 0 | 0 | 1
Menstrual disorder (Reproductive system and breast disorders) | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1
Polymenorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Uterine synechiae (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Menopausal symptoms (Reproductive system and breast disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 3 | 0 | 4
Coronary artery disease (Cardiac disorders) | 0 | 0 | 2
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 1 | 3
Dysuria (Renal and urinary disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1
Renal artery stenosis (Renal and urinary disorders) | 0 | 1 | 1
Renal colic (Renal and urinary disorders) | 0 | 0 | 1
Renal cyst (Renal and urinary disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 2
Ear congestion (Ear and labyrinth disorders) | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 2 | 0 | 1
Middle ear inflammation (Ear and labyrinth disorders) | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1
Cataract operation (Surgical and medical procedures) | 0 | 0 | 1
Hip arthroplasty (Surgical and medical procedures) | 0 | 0 | 1
Mole excision (Surgical and medical procedures) | 0 | 0 | 1
Retinal operation (Surgical and medical procedures) | 0 | 0 | 1
Rhinoplasty (Surgical and medical procedures) | 0 | 0 | 1
Tooth extraction (Surgical and medical procedures) | 0 | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic lesion (Hepatobiliary disorders) | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 1 | 1 | 5
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 2
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Blood pressure increased (Investigations) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.